CLINICAL TRIAL: NCT05764408
Title: Pannus Assistance Needed for Obstetric Ultrasound Studies: A Randomized Controlled Trial
Brief Title: Pannus Assistance Needed for Obstetric Ultrasound Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012318-1
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-07

CONDITIONS: Obesity Complicating Childbirth; Fetal Anomaly
Keywords: Obesity; Fetal ultrasound; Fetal anatomy; Pannus
MeSH Terms: conditions — Congenital Abnormalities; Obesity

STUDY DESIGN:
Masking Description: Size of varying blocks used within the permuted block design randomization will be masked to investigators. Efforts will be made to mask the physician who is interpreting the ultrasound from participant allocation; the participant and sonographer will be asked not to disclose the study arm to the interpreting physician, and no ultrasound images that would reveal study group allocation will be saved for the physician's view.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retractor (Experimental): Research team members will apply a pannus retractor adhesive according to manufacturer's directions. The sonographer will be asked to attempt all views of the detailed anatomic survey before the adhesive is removed. If the sonographer thinks that additional views could be obtained with the adhesive removed using transabdominal or transvaginal imaging, this is acceptable based on the pragmatic design of this study.
  Interventions: Device: traxi® Panniculus Retractor
- No retractor (No Intervention): The detailed anatomic survey will proceed per normal protocol. Approaches may include transabdominal and transvaginal imaging.

INTERVENTIONS:
Device: traxi® Panniculus Retractor — traxi® Panniculus Retractor is a disposable adhesive medical device designed for surgical patients with a BMI of at least 30kg/m2, to retract a pannus cephalad and expose the lower abdomen. The device is like a large sticker or bandage, posing no more than minimal risk to participants. The adhesive will be applied to the abdomen according to manufacturer instructions, just prior to a participant's scheduled ultrasound. Once the ultrasound exam has ended, the adhesive will be immediately removed and discarded.
  Arms: Retractor

SUMMARY:
The goal of this randomized controlled trial is to evaluate whether use of a pannus retractor adhesive improves fetal anatomic ultrasound examinations. The primary question it aims to answer is:

• Does the use of a pannus retractor adhesive increase the rate of detailed anatomic survey completion, defined by satisfactory visualization of sixteen prespecified fetal anatomy views, for participants with a pannus and body mass index of at least 40 kg/m2?

DETAILED DESCRIPTION:
Pregnancies complicated by obesity have an increased risk of multiple pregnancy complications, including structural fetal anomalies. Ultrasound is a critical tool for the detection of congenital anomalies; however, adequate visualization of fetal anatomy by ultrasound decreases as body mass index increases. Placing a pannus retractor adhesive is a simple intervention that redistributes adiposity, providing better access to an important acoustic window for fetal ultrasound.

The investigators will conduct a randomized controlled trial comparing outcomes between groups that undergo fetal anatomy ultrasound examinations with or without use of a pannus retractor adhesive. The adequacy of ultrasound visualization is the primary outcome of interest. Secondary outcomes of interest include sonographer pain perception, participant satisfaction, adequacy of all detailed anatomy views, detection of fetal anomalies, skin to amniotic cavity depth, duration of ultrasound exam, and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* BMI of at least 40.0 kg/2, calculated within 6 months of conception or at the first obstetric visit
* Pannus grade 1 or greater
* Gestational age between 18 weeks 0 days to 23 weeks 6 days, confirmed by prior ultrasound assessment

Exclusion Criteria:

* Patients who have already had a routinely timed anatomy ultrasound during the same pregnancy with Prisma Health Maternal-Fetal Medicine
* Patients with a known major fetal anomaly, confirmed by Prisma Health Maternal-Fetal Medicine
* Tape/adhesive allergy
* Multifetal gestation
* Intrauterine fetal demise

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pasko, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Obesity in Pregnancy: ACOG Practice Bulletin, Number 230. Obstet Gynecol. 2021 Jun 1;137(6):e128-e144. doi: 10.1097/AOG.0000000000004395. PMID 34011890
- [Background] AIUM Practice Parameter for the Performance of Detailed Second- and Third-Trimester Diagnostic Obstetric Ultrasound Examinations. J Ultrasound Med. 2019 Dec;38(12):3093-3100. doi: 10.1002/jum.15163. No abstract available. PMID 31736130
- [Background] Weichert J, Hartge DR. Obstetrical sonography in obese women: a review. J Clin Ultrasound. 2011 May;39(4):209-16. doi: 10.1002/jcu.20767. Epub 2010 Dec 7. PMID 21480286
- [Background] Dashe JS, McIntire DD, Twickler DM. Effect of maternal obesity on the ultrasound detection of anomalous fetuses. Obstet Gynecol. 2009 May;113(5):1001-1007. doi: 10.1097/AOG.0b013e3181a1d2f5. PMID 19384114
- [Background] Thornburg LL, Miles K, Ho M, Pressman EK. Fetal anatomic evaluation in the overweight and obese gravida. Ultrasound Obstet Gynecol. 2009 Jun;33(6):670-5. doi: 10.1002/uog.6401. PMID 19479682
- [Background] Bagley JE, Barnett J, Anderson MP. On-the-Job Pain and Injury as Related to Adaptive Ergonomic Equipment in the Sonographer's Workplace and Area. Journal of Diagnostic Medical Sonography, 2016. 33(1): 15-21.
- [Background] Iglesias M, Butron P, Abarca L, Perez-Monzo MF, de Rienzo-Madero B. An anthropometric classification of body contour deformities after massive weight loss. Ann Plast Surg. 2010 Aug;65(2):129-34. doi: 10.1097/SAP.0b013e3181c9c336. PMID 20606587
- [Background] Stothard KJ, Tennant PW, Bell R, Rankin J. Maternal overweight and obesity and the risk of congenital anomalies: a systematic review and meta-analysis. JAMA. 2009 Feb 11;301(6):636-50. doi: 10.1001/jama.2009.113. PMID 19211471
- [Background] Racusin D, Stevens B, Campbell G, Aagaard KM. Obesity and the risk and detection of fetal malformations. Semin Perinatol. 2012 Jun;36(3):213-21. doi: 10.1053/j.semperi.2012.05.001. PMID 22713503
- [Background] Pasko DN, Wood SL, Jenkins SM, Owen J, Harper LM. Completion and Sensitivity of the Second-Trimester Fetal Anatomic Survey in Obese Gravidas. J Ultrasound Med. 2016 Nov;35(11):2449-2457. doi: 10.7863/ultra.15.11057. Epub 2016 Oct 3. PMID 27698181
- [Background] Hendler I, Blackwell SC, Bujold E, Treadwell MC, Wolfe HM, Sokol RJ, Sorokin Y. The impact of maternal obesity on midtrimester sonographic visualization of fetal cardiac and craniospinal structures. Int J Obes Relat Metab Disord. 2004 Dec;28(12):1607-11. doi: 10.1038/sj.ijo.0802759. PMID 15303105
- [Derived] Wise ML, Okon M, Pratt KN, Lane AS, Carlson LM, Eichelberger KY, Crockett AH, Zhang L, Pasko DN. Panniculus Retractor Use for Visualization of Fetal Anatomy: A Randomized Controlled Trial. Obstet Gynecol. 2024 Sep 1;144(3):403-410. doi: 10.1097/AOG.0000000000005689. Epub 2024 Jul 25. PMID 39053011

RESULTS

PARTICIPANT FLOW:
Groups:
- Retractor: Anatomy ultrasound performed with panniculus retractor
- Control: Anatomy ultrasound performed through usual protocol without a retractor
Period: Overall Study
Arm/Group | Retractor | Control
Started | 74 | 76
Completed | 74 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retractor | Control | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (5.27) | 28.9 (4.63) | 28.6 (4.95)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Pregnant | 74 | 76 | 150
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Insurance status [Count of Participants; unit: Participants]
  Private | 32 | 28 | 60
  Public | 37 | 36 | 73
  Private and public | 3 | 8 | 11
  Other | 1 | 0 | 1
  None | 1 | 4 | 5
Tobacco use [Count of Participants; unit: Participants] | 5 | 7 | 12
Diabetes mellitus [Count of Participants; unit: Participants]
  Pregestational | 4 | 7 | 11
  Gestational | 8 | 5 | 13
  None | 62 | 64 | 126
Prior cesarean delivery [Count of Participants; unit: Participants]
  Yes | 27 | 18 | 45
  No | 47 | 58 | 105
Other abdominal surgery [Count of Participants; unit: Participants]
  Yes | 23 | 15 | 38
  No | 51 | 61 | 112
Nulliparous [Count of Participants; unit: Participants]
  Yes | 19 | 23 | 42
  No | 55 | 53 | 108
Cephalic presentation [Count of Participants; unit: Participants]
  Yes | 30 | 33 | 63
  No | 44 | 43 | 87
Gestational age at ultrasound, weeks [Mean (Standard Deviation); unit: Weeks] | 20.6 (0.72) | 20.4 (0.74) | 20.5 (0.73)
Waist circumference, inches [Mean (Standard Deviation); unit: inches] | 56.8 (5.20) | 56.4 (4.41) | 56.6 (4.81)
Body mass index, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 46.7 (5.04) | 46.2 (5.00) | 46.5 (5.02)
Panniculus grade [Count of Participants; unit: Participants] — Panniculus grade was evaluated in a reclined, supine position. It was classified according to the system described by Iglesias et al.: no panniculus (grade 0), panniculus remaining above the inguinal ligament (grade 1), overhanging panniculus below the inguinal ligament but not surpassing the upper third of the thigh (grade 2), overhanging panniculus located within the middle third of the thigh (grade 3), overhanging panniculus within the lower third of the thigh (grade 4), overhanging panniculus below the knee (grade 5). Higher grades indicate a more significant panniculus presence.
  Participants
    1 | 34 | 50 | 84
    2 | 38 | 23 | 61
    3 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate of 16 Prespecified Views
Description: Views including: brain (lateral ventricles, cerebellum, cavum), face, heart (four chamber view, right outflow tract, left outflow tract, three vessel view, three vessel trachea view), spine (cervical, thoracic, lumbar, sacrum, and spine shape will be summarized as one spine view), ventral wall, umbilical cord, stomach, left and right kidneys, and bladder.
Time Frame: through study completion, an average of 1 day per participant
Measure: Count of Participants; unit: Participants
Arm/Group | Retractor | Control
Number analyzed (Participants) | 74 | 76
Participants | 19 | 24
Statistical Analysis 1: Comparison: Retractor vs Control; Test type: Superiority; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.49 to 1.35]

2. Secondary Outcome: Completion Rate of All 64 Views
Description: Views including: calvarium/cranium, intracranial anatomy, cavum, parenchyma, lateral ventricles, choroid plexus, cerebellum/vermis, cisterna magna, midline falx, cervical spine, thoracic spine, lumbar spine, sacral spine, spine shape/curvature, face, lips, neck, nuchal fold, nasal bone, palate, profile, orbits/eyes, mandible, maxilla, thoracic contour, lungs, four chamber view, cardiac activity, cardiac rhythm, cardiac situs, right outflow tract, left outflow tract, aortic arch, ductal arch, SVC, interventricular septum, cardiac axis, diaphragm, three vessel view, three vessel trachea view, IVC, crossing, ventral wall, cord insertion, situs, stomach, gallbladder, left kidney, right kidney, bladder, left humerus, right humerus, left forearm, right forearm, left hand, right hand, left femur, right femur, left lower leg, right lower leg, left foot, right foot, umbilical cord, genitalia.
Time Frame: through study completion, an average of 1 day per participant
Measure: Count of Participants; unit: Participants
Arm/Group | Retractor | Control
Number analyzed (Participants) | 74 | 76
Participants | 10 | 12
Statistical Analysis 1: Comparison: Retractor vs Control; Test type: Superiority; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.39 to 1.86]

3. Secondary Outcome: Duration of Ultrasound Exam
Description: The time from first to last ultrasound image acquisition, time for retractor placement not included
Time Frame: through study completion, an average of 1 day per participant
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Retractor | Control
Number analyzed (Participants) | 74 | 76
minutes | 34.9 (10.46) | 33.7 (11.24)
Statistical Analysis 1: Comparison: Retractor vs Control; Test type: Superiority; p = 0.47, t-test, 2 sided

4. Secondary Outcome: Detection of Major Fetal Anomalies
Description: Per EUROCAT guidelines
Time Frame: through study completion, an average of 1 day per participant
Measure: Count of Participants; unit: Participants
Arm/Group | Retractor | Control
Number analyzed (Participants) | 74 | 76
Participants | 0 | 0

5. Secondary Outcome: Depth to Amniotic Cavity
Description: Using only the minimal amount of pressure to create the image, the shortest mid-sagittal distance will be measured from the skin to the amniotic cavity above and below the panniculus. This is for the retractor group only.
Time Frame: through study completion, an average of 1 day per participant
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Retractor
Number analyzed (Participants) | 74
centimeters
  Before retractor | 5.0 (1.64)
  After retractor | 5.0 (1.71)
Statistical Analysis 1: Comparison: Retractor; Test type: Superiority; p = 0.81, t-test, 2 sided

6. Secondary Outcome: Adverse Effects
Description: In addition to routine monitoring for all adverse effects, the following will be noted specifically: skin irritation, allergic reaction, maternal intolerance of pannus retractor adhesive, fetal demise, and hospital admission immediately following the ultrasound exam.
Time Frame: through study completion, an average of 1 day per participant
Measure: Count of Participants; unit: Participants
Arm/Group | Retractor | Control
Number analyzed (Participants) | 74 | 76
Participants
  Skin irritation | 0 | 1
  Allergic reaction | 0 | 0
  Fetal demise | 0 | 0
  Hospital admission | 1 | 0
  None | 73 | 75
Statistical Analysis 1: Comparison: Retractor vs Control; Test type: Superiority; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.07 to 16.12]

7. Secondary Outcome: Sonographer Survey
Description: Immediately after the ultrasound exam, a survey was administered to the sonographer who performed the anatomy ultrasound for each participant. The questions were asked with Likert scale responses ranging from strongly disagree (1) to strongly agree (5).
Time Frame: through study completion, an average of 1 day per participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retractor | Control
Number analyzed (Participants) | 74 | 76
score on a scale
  I experienced pain in my arm, shoulder, and/or wrist while performing this ultrasound | 3.7 (1.21) | 3.9 (1.03)
  The participant's body habits affected my ability to complete the ultrasound | 4.1 (1.05) | 4.3 (0.94)
  I feel confident about the quality of ultrasound images obtained | 3.8 (0.99) | 3.6 (0.98)

8. Secondary Outcome: Participant Survey
Description: Immediately after the ultrasound exam, a survey was administered to the participant. The questions were asked with Likert scale responses ranging from strongly disagree (1) to strongly agree (5).
Time Frame: through study completion, an average of 1 day per participant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Retractor | Control
Number analyzed (Participants) | 74 | 76
score on a scale
  I felt comfortable during the ultrasound | 4.6 (0.84) | 4.8 (0.44)
  I am satisfied with the quality of ultrasound pictures I received | 4.6 (0.70) | 4.5 (0.60)
  I enjoyed the ultrasound experience today | 4.6 (0.69) | 4.7 (0.52)

ADVERSE EVENTS:
Time Frame: Same day as ultrasound
Arm/Group | Retractor | Control
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/74 | 0/76
Other Adverse Events (participants affected / at risk) | 0/74 | 1/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retractor (N=74) | Control (N=76)
Hospital admission (Social circumstances) | 1 | 0 — Hospital admission following the ultrasound examination was collected for any medical reason. The one admission seen was for cervical insufficiency unrelated to the trial.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retractor (N=74) | Control (N=76)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT05764408/Prot_SAP_000.pdf